CLINICAL TRIAL: NCT02326480
Title: Genetic Analysis of Childhood Obesity
Acronym: OSV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Collaborators: Institut Pasteur de Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0036
Record Dates: First submitted 2014-12-15; First posted 2014-12-29 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Obesity
Keywords: Childhood Obesity; Genetics
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Syndromic obesity: Identification of genetic causes of obesity
- Familial obesity: Identification of genetic causes of obesity
  Interventions: Other: Identification of genetic causes of obesity
- Isolated obesity: Identification of genetic causes of obesity
  Interventions: Other: Identification of genetic causes of obesity

INTERVENTIONS:
Other: Identification of genetic causes of obesity — A blood test will be performed to the child and his/her parents with the aim of identifying genetic causes of obesity. Different analysis will be as follows: caryotypes, Raindance, whole exome, in order to find potential mutations or new genes associated to this condition
  Groups: Familial obesity; Isolated obesity

SUMMARY:
Identify news genetic causes of different type of obesity (syndromic, familial or isolated obesity) by highlighting new mutations or new implied genes

ELIGIBILITY:
Inclusion criteria:

* BMI > curve of IOTF 30 (International Obesity Task Force)
* Age: between 6 months old and 18 years old
* Child presenting syndromic, isolated or familial obesity.

Exclusion Criteria:

* Common obesity
* Impossibility for blood sampling
* Impossibility to receive information
* Participation refusal of one of the parents
* Refusal to sign the informed consent
* Neither Healthcare coverage nor insurance

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Three categories of obese children with their biological parents will be included (syndromic, familial, isolated obesity).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
To identify the number of mutations or genes involved in genetic causes of Child obesity | first day of enrollement
  Children with obesity and their parents will be recruited to establish genetic causes of obesity. This will allow perform genetic analysis using new approaches for the identification of involved mutations or new candidate genes

SECONDARY OUTCOMES:
To identify the number of mutations in the population | first day of enrollement
To identify the number of new mutations present in the children's DNA and absent from their parents' genomes | first day of enrollement
  This approach will allow the identification of specific mutations that are present only in affected children but not in their parents
To determine number of phenotypes associated to the child obesity genotype | first day of enrollement

CONTACTS AND LOCATIONS:
Overall Officials: Louise Montagne, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille; Philippe Froguel, MD, PhD, Principal Investigator — UMR CNRS 8199, Institut Pasteur de Lille
Locations (1):
- Hôpital Saint Vincent de Paul, Lille, France